CLINICAL TRIAL: NCT03064620
Title: PICR-b Nasopharyngeal S. Pneumoniae and Nasal S. Aureus Carriage Study
Acronym: PICRcarriage
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Palestinian-Israeli Collaborative Research (PICR) (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); The Israeli National Institute for Health Policy Research (Unknown); Maccabi Healthcare Services, Israel (Other)
Responsible Party: Principal Investigator, Gili Regev-Yochay MD, Head of Infect Dis Epi Section, Gertner, Sheba Medical Center
Other Study IDs: 8024-10
Record Dates: First submitted 2016-03-29; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Streptococcus Pneumoniae
Keywords: PCV effects; S. pneumoniae carriage; S. aureus carriage; Indirect vaccination effects; Palestinian-Israeli Collaborative Research (PICR)
MeSH Terms: interventions — 10-valent pneumococcal conjugate vaccine

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — S. aureus and S. pneumoniae
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Israel PCV13: Children and their parents living in central Israel and visiting primary pediatric clinics of Hashfela District, Macabbi Healthcare Services HMO, for any reason during the surveillance period each year.
  Interventions: Biological: PCV
- East Jerusalem PCV13: Children and their parents living in East Jerusalem and visiting primary pediatric clinics of Jerusalem District, Macabbi Healthcare Services HMO, for any reason during the surveillance period each year.
  Interventions: Biological: PCV
- Palestine PCV7 PCV10: Children and their parents living in major cities of the Palestinian Authority and visiting private primary pediatric clinics, for any reason during the surveillance period each year.
  Interventions: Biological: PCV

INTERVENTIONS:
Biological: PCV — PCV7 was introduced in Israel (IL and EJ) in July 2009 PCV13 replaced PCV7 in IL and EJ on Oct 2010 PCV10 was introduced in PA in 2011
  Other Names: PCV7; PCV10; PCV13

SUMMARY:
Objective: PCV effects on S. pneumoniae and S. aureus carriage in a population based study. The major specific aims:

1. To compare different PCV vaccination policies, by cross-sectional repeated surveillance of closely related populations living in regions with different vaccination policies.
2. To compare the epidemiology, predictors and outcomes of antibiotic resistant S. aureus and S. pneumoniae in different regions of the PICR.

Study design: Annual / Biannual cross-sectional surveillance of nasal S. aureus carriage and nasopharyngeal S. pneumoniae carriage in children and one of their parents.

DETAILED DESCRIPTION:
Study design: Annual / Biannual cross-sectional surveillance of nasal S. aureus carriage and nasopharyngeal S. pneumoniae carriage in children and one of their parents.

PICR districts: 1. Palestinian Authority (PA) - particularly: Bethlehem, Ramallah and Nabulus. 2. East Jerusalem (EJ) 3. Central Israel (IL) - particularly: Rishon Lezion, Bat Yam, Holon 4. Gaza strip (GZ) - 12 regions including cities/villages in central/northern Gaza.

Study population:

Child (age 0-5y) & Parent who attend clinics (for any reason).

Exclusion criteria:

Parent does not agree to sign informed consent Child or sibling (brother/sister) have already participated.

Both healthy and ill children are screened. No specific exclusion other than the above.

Only one child per family (younger child, if more than one available) and one parent (mother, if both are available).

Sample size per year:

IL: Central Israel (Hashfela District): 400 pairs of child+parent/surveillance EJ: East Jerusalem: 400 pairs of child+parent/surveillance PA: West Bank cities (Ramallah, Bethlehem & Nabulus): 600 pairs of child+parent/surveillance GZ: Gaza strip: 300 pairs of child+parent/surveillance

Study Period:

May-August annually 2009 - 2011 - (Part a). May-August biannually 2014-2016-2018-2020 Current study (Part b).

Screening Procedure:

1. Parent signs informed consent
2. Put Barcode stickers on informed consent, questionnaire, swabs and daily list
3. Fill questionnaire with parent.
4. Fill physician questionnaire
5. Nasal & nasopharyngeal swab of child and parent.
6. Fill daily working table.
7. Write the number of refusals (parents who refused) on daily table.
8. Fill questionnaire FULLY (unmarked questions will not be analyzed) - put x on each question - whether YES or NO.

Swabbing:

1. First swab the child and then follow with the parent.
2. First perform nasal swab (for S. aureus) using cotton-tip swab placed into Amies transport Media (Blue) and follow with nasopharyngeal swab ( for S. pneumoniae) using rayon-tipped aluminum shaft swab placed in Amies transport Media (Orange).
3. Slightly wet the nasal swab with sterile saline. Swab both anterior nares.
4. Nasopharyngeal swab of only through one nostril - gently, quickly and deep to nasopharynx - until you touch the nasopharyngeal wall.

Swab transfer to lab:

If swabs are stored overnight before transfer - keep in 40C (fridge). Within 24h swabs must reach the central laboratory (Dr. Regev-Yochay's Lab at Sheba Medical Center).

ELIGIBILITY:
Inclusion Criteria:

* Any child younger than 5 years, visiting the participating clinics during the surveillance period

Exclusion Criteria:

* Older than 5 years
* Previously participated in the study.
* Sibling has participated in the study.
* Parent does not agree to sign informed consent

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Child (age 0-5y) & Parent who attend pediatric clinics (for any reason), in the participating clinics during the surveillance periods.
Sampling Method: Probability Sample
Enrollment: 12800 (Estimated)
Dates: Start 2014-04; Primary Completion 2020-08 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
S. pneumoniae carriage | 1 Day
  S. pneumoniae carriage of children and parents by the different groups

SECONDARY OUTCOMES:
Carriage of Vaccine-type S. pneumoniae | 1 Day
  Carriage of Vaccine-type S. pneumoniae in children and parents by the different groups
Carriage of antibiotic resistant S. pneumonia | 1 Day
  Carriage of antibiotic resistant S. pneumonia in children and parents by the different groups
Carriage of piliated S. pneumonia | 1 Day
  Carriage of piliated S. pneumonia in children and parents by the different groups
Carriage of MRSA | 1 Day
  Carriage of MRSA in children and parents by the different groups
S. aureus carriage | 1 Day
  S. aureus carriage of children and parents by the different groups

CONTACTS AND LOCATIONS:
Overall Officials: Dror Harats, Prof., Study Chair — IRB Committee Sheba Medical Center Israel
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daana M, Rahav G, Hamdan A, Thalji A, Jaar F, Abdeen Z, Jaber H, Goral A, Huppert A, Raz M, Regev-Yochay G; PICR study group. Measuring the effects of pneumococcal conjugate vaccine (PCV7) on Streptococcus pneumoniae carriage and antibiotic resistance: the Palestinian-Israeli Collaborative Research (PICR). Vaccine. 2015 Feb 18;33(8):1021-6. doi: 10.1016/j.vaccine.2015.01.003. Epub 2015 Jan 12. PMID 25593104
- [Background] Southern J, Roizin H, Daana M, Rubin C, Hasleton S, Cohen A, Goral A, Rahav G, Raz M, Regev-Yochay G; PICR group. Varied utilisation of health provision by Arab and Jewish residents in Israel. Int J Equity Health. 2015 Aug 7;14:63. doi: 10.1186/s12939-015-0193-8. PMID 26245327
- [Background] Regev-Yochay G, Abullaish I, Malley R, Shainberg B, Varon M, Roytman Y, Ziv A, Goral A, Elhamdany A, Rahav G, Raz M; Palestinian-Israeli Collaborative Research Study Group. Streptococcus pneumoniae carriage in the Gaza strip. PLoS One. 2012;7(4):e35061. doi: 10.1371/journal.pone.0035061. Epub 2012 Apr 23. PMID 22539955
- [Background] Biber A, Abuelaish I, Rahav G, Raz M, Cohen L, Valinsky L, Taran D, Goral A, Elhamdany A, Regev-Yochay G; PICR Study Group. A typical hospital-acquired methicillin-resistant Staphylococcus aureus clone is widespread in the community in the Gaza strip. PLoS One. 2012;7(8):e42864. doi: 10.1371/journal.pone.0042864. Epub 2012 Aug 16. PMID 22916171